CLINICAL TRIAL: NCT00003143
Title: A Randomized Study of Ethyol (Amifostine) With Platinum Based Salvage Chemotherapy in Patients With Lymphoma Undergoing Autologous Stem Cell Transplantation
Brief Title: Combination Chemotherapy With or Without Amifostine in Treating Patients With Recurrent or Refractory Non-Hodgkin's Lymphoma or Hodgkin's Disease Undergoing Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000065926; UCLA-HSPC-970708701; ALZA-UCLA-HSPC-970708701; NCI-V97-1362
Record Dates: First submitted 1999-11-01; First posted 2004-06-16 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma; Waldenström macroglobulinemia; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Waldenstrom Macroglobulinemia; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Amifostine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DHAP + amifostine (Experimental): Patients are randomized to receive salvage chemotherapy with intravenous dexamethasone/cisplatin/cytarabine (DHAP) with or without amifostine. Patients receive cisplatin IV over 3 hours followed by cytarabine IV for 2 doses. Patients also receive dexamethasone orally or IV. Treatment repeats every 3-4 weeks for 2-6 courses. Arm I: Patients receive amifostine IV over 15 minutes prior to all courses of DHAP, as a 15 minute infusion, beginning 30 minutes prior to cisplatin administration. Arm II: Patients do not receive amifostine. On day 3 of the last DHAP course, patients receive filgrastim (G-CSF) until the last day of progenitor stem cell (PSC) mobilization. PSC transplant continues daily for 4-10 days.
  Interventions: Drug: Amifostine; Drug: DHAP
- DHAP (Other): Patients are randomized to receive salvage chemotherapy with intravenous dexamethasone/cisplatin/cytarabine (DHAP) with or without amifostine. Patients receive cisplatin IV over 3 hours followed by cytarabine IV for 2 doses. Patients also receive dexamethasone orally or IV. Treatment repeats every 3-4 weeks for 2-6 courses. Arm I: Patients receive amifostine IV over 15 minutes prior to all courses of DHAP, as a 15 minute infusion, beginning 30 minutes prior to cisplatin administration. Arm II: Patients do not receive amifostine. On day 3 of the last DHAP course, patients receive filgrastim (G-CSF) until the last day of progenitor stem cell (PSC) mobilization. PSC transplant continues daily for 4-10 days.
  Interventions: Drug: DHAP

INTERVENTIONS:
Drug: Amifostine
  Arms: DHAP + amifostine
Drug: DHAP

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Chemoprotective drugs such as amifostine may protect normal cells from the side effects of chemotherapy.

PURPOSE: Randomized phase II trial to study the effectiveness of combination chemotherapy with or without amifostine in treating patients with recurrent or refractory non-Hodgkin's lymphoma or Hodgkin's disease who are undergoing autologous stem cell transplantation.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the role of amifostine in reducing hematologic toxicity and improving mobilization of peripheral progenitor stem cells in patients with recurrent or refractory non-Hodgkin's lymphoma or Hodgkin's disease who are undergoing platinum based salvage chemotherapy. II. Evaluate the role of amifostine in preventing renal toxicity in these patients.

OUTLINE: This is an randomized, open label study. Patients are randomized to receive salvage chemotherapy with intravenous dexamethasone/cisplatin/cytarabine (DHAP) with or without amifostine. Patients receive cisplatin IV over 3 hours followed by cytarabine IV for 2 doses. Patients also receive dexamethasone orally or IV. Treatment repeats every 3-4 weeks for 2-6 courses. Arm I: Patients receive amifostine IV over 15 minutes prior to all courses of DHAP, as a 15 minute infusion, beginning 30 minutes prior to cisplatin administration. Arm II: Patients do not receive amifostine. On day 3 of the last DHAP course, patients receive filgrastim (G-CSF) until the last day of progenitor stem cell (PSC) mobilization. PSC transplant continues daily for 4-10 days.

PROJECTED ACCRUAL: A total of 40 patients (20 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven recurrent or refractory non-Hodgkin's lymphoma or Hodgkin's disease requiring salvage chemotherapy Prior treatment with at least 3 courses of first line chemotherapy

PATIENT CHARACTERISTICS: Age: Over 18 Performance Status: ECOG 0-2 Life Expectancy: Greater than 3 months Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 50,000/mm3 Hepatic: Not specified Renal: Creatinine no greater than 1.5 mg/dL Creatinine clearance at least 40 mL/min Cardiovascular: No symptomatic congestive heart failure (class III or more as defined by American Heart Association) Electrolytes: Potassium at least 3.4 meq/L Magnesium at least 1.4 meq/L Other: Not pregnant or nursing

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior high dose chemotherapy with stem cell transplant At least 3 courses of first line chemotherapy Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 1997-11; Primary Completion 2000-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christos E. Emmanouilides, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States